CLINICAL TRIAL: NCT04246190
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety After Oral Administration of CKD-396 and Co-administration of CKD-501 and D759 in Healthy Adults
Brief Title: A Clinical Study to Evaluate the Pharmacokinetics and Safety of CKD-396
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A65_03BE1921
Record Dates: First submitted 2020-01-28; First posted 2020-01-29 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — lobeglitazone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): * Period 1: CKD-501 and D759
  * Period 2: CKD-396
  Interventions: Drug: CKD-501 and D759; Drug: CKD-396
- Group 2 (Experimental): * Period 1: CKD-396
  * Period 2: CKD-501 and D759
  Interventions: Drug: CKD-501 and D759; Drug: CKD-396

INTERVENTIONS:
Drug: CKD-501 and D759 — Reference drug, CKD-501 1T and D759 1T, QD, PO
Drug: CKD-396 — Reference drug, CKD-396 1T, QD, PO

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of CKD-396.

DETAILED DESCRIPTION:
Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety After Oral Administration of CKD-396 and Co-administration of CKD-501 and D759 in Healthy Adults

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult who is 19 ~ 55 years at the time of screening
2. Body weight more than 55 kg for male and more than 50kg for female
3. BMI more than 18.5 kg/m2 or less than 27.0 kg/m2
4. Females must be menopause or surgical infertility
5. Males who have consented to the use of appropriate pregnancy contraceptive methods up to 28 days after the last investigational product and not to provide sperm
6. Subjects who voluntarily decided to participate and informed consent based upon understanding on the study.

Exclusion Criteria:

1. Subjects who have a history of clinically significant hepatic, renal, nervous, immune, respiratory, urinary, digestion, endocrine, hematooncology, cardiovascular systemic disease or psychosis disorder
2. Subjects who have diabetic ketoacidoisis, diabetic coma, diabetic precoma, Type 1 diabetes
3. Subjects who have genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
4. Subjects who have a history of gastrointestinal disorders (Crohn's disease, ulcerative colitis, etc.) or surgery (except simple appendectomy or hernia surgery) that may affect the absorption of the drug
5. Subjects who have a history of clinically significant hypersensitivity to drugs or additives, including components of the investigational product(lobeglitazone, sitagliptin) and same class drug with thiazolidinediones
6. Subjects who have severe infectious disease and severe trauma before and after operation
7. Subjects who are deemed unsuitable as subjects in the screening test performed within 28 days before the administration of investigational product

   * AST, ALT> UNL(Upper Normal Limit)x1.25
   * Total bilirubin > UNL(Upper Normal Limit)x1.5
   * eGFR (Estimated Glomerular Filtration Rate) <60 mL/min/1.73m2 using the MDRD (Modification of Diet in Renal Disease) formula
   * Positive immunologic serological tests (hepatitis B test, hepatitis C test, human immunodeficiency virus (HIV) test, syphilis test)
   * After resting for more than 5 minutes, systolic blood pressure> 150 mmHg or < 90 mmHg, diastolic blood pressure> 100 mmHg or <50 mmHg
8. Subjects who have had a history of drug abuse within one year of screening or have tested positive on urine drug screening test
9. Pregnant or lactating women
10. Subjects who have consistently excessively smoked or consumed caffeine or alcohol (caffeine:> 5 cups / day, alcohol:> 210 g / week, cigarettes:> 10 cigarettes / day) or cannot stop smoking, consuming caffeine and alcohol during hospitalization
11. Subjects who judged to able to affect in the study or in the subject's safety by the investigator for the following reasons

    * Ethical-the-counter (ETC) drugs and herbal medicines within 14 days of the first administration of the investigational drug.
    * Over-the-counter (OTC) drugs, including health foods and vitamin preparations, within 7 days of the first dose of the investigational product
12. Subjects who have received the investigational product by participating in other clinical trials (including bioequivalence studies) within 180 days before the first dose of the investigational product (For biological agents, this may be based on a longer period of time, considering the half-life)
13. Subjects who donated whole blood within 60 days before the first dose of the investigational product or donated component blood donation within 30 days
14. Subjects who received a blood transfusion within 60 days before the first dose of the investigational product
15. Subjects who were deemed to be inappropriate to participate in the study by the investigator judgment

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-02-24 (Estimated); Primary Completion 2020-04-10 (Estimated); Study Completion 2020-07-16 (Estimated)

PRIMARY OUTCOMES:
Cmax of CKD-501, D759 and CKD-396 | 0(predose)~48 hours
  Maximum plasma concentration of CKD-501, D759 and CKD-396
AUClast of CKD-501, D759 and CKD-396 | 0(predose)~48 hours
  Area under the plasma concentration-time curve to last concentration of CKD-501, D759 and CKD-396

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, Ph.D. M.D, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Severance Hospital, Soeul, South Korea